CLINICAL TRIAL: NCT03931005
Title: Collaborating to Implement Cross-System Interventions in Child Welfare and Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017B0239
Record Dates: First submitted 2019-04-22; First posted 2019-04-29 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-02

CONDITIONS: Substance Use; Implementation; Child Maltreatment; System Fragmentation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision-Support (Experimental): An electronic copy of a collaboration decision-support guide.
  Interventions: Other: Collaboration Decision Support Guide

INTERVENTIONS:
Other: Collaboration Decision Support Guide — Electronic toolkit intended to help organizational leaders select partners and negotiate partnerships for implementation. This will contain: 1) a brief summary of collaboration approaches associated with implementation, 2) detailed descriptions of collaboration strategies, 3) a decision analysis tool that guides the selection of collaborative strategies given the community context, and 4) sample contract or agreement language that specifies the nature of the partnership and expectations.

SUMMARY:
As a result of the opiate crisis, child welfare agencies have experienced an increase in the number of children in foster care as parental substance use puts children at greater risk of maltreatment. To facilitate implementation of the Sobriety Treatment and Recovery Team (START) model, this study (1) identifies collaborative strategies associated with effective implementation and service outcomes given system and organizational context, (2) uses this evidence to specify strategies and develop a decision support guide to help agency leaders select collaborative strategies, and (3) assesses the feasibility, acceptability, and appropriateness of the decision support guide.

DETAILED DESCRIPTION:
This is a multi-staged, mixed methods study that leverages a naturally occurring policy experiment in southern Ohio. In aim 1, we will examine the collaborative strategies associated with implementation and service outcomes, given the context with 17 counties engaged in the Ohio START pilot project. We will use a convergent mixed methods design, and integrate our qualitative and quantitative data using qualitative comparative analysis. For aim 2, we will specify the collaborative strategies and develop a decision support guide using the VA's model of implementation strategy development (diagnose barriers, and convene an expert panel to design strategies). For aim 3, we assess the feasibility, acceptability, and appropriateness of the decision support guide using a sequential mixed methods design. In the first quantitative phase, we will conduct a randomized vignette experiment with agency directors in the 71 Ohio counties that are not involved in the Ohio START pilot project to compare the decision support guide with general implementation support. Our second qualitative phase (which is dominant), will examine feasibility more in-depth by piloting the guide and conducting descriptive case studies with up to three new counties.

ELIGIBILITY:
Inclusion Criteria:

* Our participants included implementation support professionals who provide training and technical assistance to child welfare agencies in Ohio that are implementing Ohio START. All individuals will be adults and recruited based on their employment/position.

Exclusion Criteria:

* Individuals who do not provide implementation support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Perceived Acceptability | One time point (Post-test only), immediately after receipt of intervention
  Acceptability of Intervention Measure (AIM) - 4 survey items that assess participants' agreement about the degree to which they perceive the intervention to be acceptable. Participants rate their agreement along a 5 point scale, where 1= completely disagree and 5= completely agree. Scores from the four items will be averaged where higher scores denote greater perceived acceptability. (Weiner, B. J., Lewis, C. C., Stanick, C., Powell, B. J., Dorsey, C. N., Clary, A. S., … Halko, H. (2017). Psychometric assessment of three newly developed implementation outcome measures. Implementation Science, 12(108), 1-12. https://doi.org/10.1186/s13012-017-0635-3)
Perceived Appropriateness | One time point (Post-test only), immediately after receipt of intervention
  Intervention Appropriateness Measure (IAM) - 4 survey items that assess participants' agreement about the degree to which they perceive the intervention to be appropriate. Participants rate their agreement along a 5 point scale, where 1= completely disagree and 5= completely agree. Scores from the four items will be averaged where higher scores denote greater perceived appropriateness. (Weiner, B. J., Lewis, C. C., Stanick, C., Powell, B. J., Dorsey, C. N., Clary, A. S., … Halko, H. (2017). Psychometric assessment of three newly developed implementation outcome measures. Implementation Science, 12(108), 1-12. https://doi.org/10.1186/s13012-017-0635-3)
Perceived Feasibility | One time point (Post-test only), immediately after receipt of intervention
  Feasibility of Intervention Measure (FIM) - 4 survey items that assess participants' agreement about the degree to which they perceive the intervention to be feasible. Participants rate their agreement along a 5 point scale, where 1= completely disagree and 5= completely agree. Scores from the four items will be averaged where higher scores denote greater perceived feasibility. (Weiner, B. J., Lewis, C. C., Stanick, C., Powell, B. J., Dorsey, C. N., Clary, A. S., … Halko, H. (2017). Psychometric assessment of three newly developed implementation outcome measures. Implementation Science, 12(108), 1-12. https://doi.org/10.1186/s13012-017-0635-3)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Bunger, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chuang E, Bunger A, Smith R, Girth A, Phillips R, Miech E, Lancaster K, Martin J, Gadel F, Himmeger M, McClellan J, Millisor J, Willauer T, Powell BJ, Dellor E, Aarons GA. Collaboration strategies affecting implementation of a cross-systems intervention for child welfare and substance use treatment: a mixed methods analysis. Implement Sci Commun. 2024 Nov 11;5(1):127. doi: 10.1186/s43058-024-00666-w. PMID 39529175
- [Derived] Bunger AC, Chuang E, Girth A, Lancaster KE, Gadel F, Himmeger M, Saldana L, Powell BJ, Aarons GA. Establishing cross-systems collaborations for implementation: protocol for a longitudinal mixed methods study. Implement Sci. 2020 Jul 16;15(1):55. doi: 10.1186/s13012-020-01016-9. PMID 32677987